CLINICAL TRIAL: NCT07226050
Title: A Randomized, Placebo-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of CLF065 in the Treatment of Chronic Pouchitis
Brief Title: CLF065 for Chronic Pouchitis
Acronym: OPUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBR-CLF065-4001
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pouchitis
Keywords: chronic pouchitis
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLF065 (Experimental): CLF065 subcutaneous weekly
  Interventions: Drug: CLF065
- Placebo (Placebo Comparator): Matching placebo subcutaneous weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLF065 — will receive investigational product every week for 13 weeks as a sub-cutaneous injection
  Arms: CLF065
Drug: Placebo — CLF065 matching placebo
  Arms: Placebo

SUMMARY:
This clinical trial is to evaluate investigational compound CLF065 as a treatment for adult patients with chronic pouchitis. The goals are to establish the safety, feasibility and efficacy of weekly dosing of long acting CLF065 versus placebo.

DETAILED DESCRIPTION:
CLF065 is a long acting Glucagon-like peptide-2 (GLP-2). Participants will receive CLF065 or a placebo as a subcutaneous injection (just under the skin) once a week for the first 13 weeks of a 24-week total study period. Some weeks the subcutaneous injection will be given at the study site and some weeks it will be self-administered. Participants will be asked to complete a daily bowel diary card in addition to questionnaires about living with chronic pouchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18-80 years, inclusive.
2. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
3. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
4. Diagnosis of pouchitis that is recurrent, defined by mPDAI score of > 5 assessed as the average from 3 days immediately prior to Baseline endoscopy, and a minimum endoscopic subscore of 2 (outside the staple or suture line) with either:

   > 3 episodes of pouchitis within 1 year of Screening visit, each treated with antibiotic or other prescription therapy for at least 2 weeks OR Requiring maintenance antibiotic therapy taken continuously for >4 weeks immediately prior to the Baseline endoscopic visit
5. The patient has a history of proctocolectomy and construction of an IPAA for ulcerative colitis at least one year before the Screening Visit.
6. The patient agrees to stop antibiotic therapy on Day 1 of the study.
7. Patient agrees to taper any corticosteroid or budesonide starting by Week 4 of the study per guidelines below.
8. A male subject who is nonsterilized and sexually activity with a female partner of childbearing potential agrees to use a barrier method of contraception (e.g., condom with spermicide) from signing informed consent throughout the duration of the study.
9. Women of childbearing potential must not have a positive pregnancy test at the Screening Visit and must have a negative pregnancy test at the baseline visit prior to study drug dosing. Note: subjects with borderline serum pregnancy test at Screening must have an absence of clinical suspicion of pregnancy or other pathological cause of a borderline result and a serum pregnancy test ≥ 3 days later to document continued lack of a positive result.
10. If female, the patient must be either postmenopausal, OR permanently surgically sterile or for women of childbearing potential practicing at least one protocol specified method of birth control, that is effective from baseline visit through at least 30 days after the last dose of study drug.
11. Patient is judged to be in good health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination

Exclusion Criteria:

1. Inability to give informed consent.
2. The patient has received any investigational product or approved biologic or biosimilar agent within 60 days of 5 half-lives of randomization (whichever is longer)
3. No prior exposure to CLF065
4. Chronic pouchitis specific:

   1. The patient has received 6-MP, Azathioprine or methotrexate within 4 weeks of the Screening Visit
   2. Crohn's disease with disease proximal to the pouch inlet confirmed on prior imaging or endoscopy
   3. Irritable pouch syndrome
   4. Predominate or isolated cuffitis
   5. Mechanical complications of the pouch
   6. Diverting stoma
   7. Planned surgical intervention of the pouch
5. History of malignancy including melanoma (with the exception of localized skin cancers, carcinoma in situ of the cervix and localized prostate cancer) within 2 years of study enrollment
6. Pregnant or breast feeding.
7. Lack of effective contraception in women of childbearing potential.
8. Ongoing treatment with NSAID (nonsteroidal anti-inflammatory drug).
9. Anastomotic or anal canal stricture which precludes endoscopic evaluation.
10. The patient has evidence of pelvic sepsis and pelvic penetrating fistulizing disease on clinical exam.
11. Known diagnosis of primary sclerosing cholangitis.
12. Fecal transplantation within 12 weeks prior to study enrollment.
13. History of clinically significant medical conditions or any other reason that in the opinion of the investigator would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study drug or would put the subject at risk by participating in the study.
14. The patient has any of the following laboratory abnormalities during the Screening Period:

    1. Hemoglobin level <8 g/dL
    2. White blood cell (WBC) count <3 x 109/L
    3. Platelet count <100 x 109/L or >1200 x 109/L
    4. Serum creatinine >2 x ULN
    5. Alanine aminotransferase (ALT) or aspartate aminiotransferase (AST) >3x ULN
    6. Alkaline phosphatase >3 x ULN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Pouchitis Disease Activity Index (PDAI) and Modified PDAI | Baseline, Week 14, Week 24
  The PDAI contains three separate 6-point domain scales based on clinical symptoms, endoscopic inflammation, and acute histologic inflammation. On the scale, 0 = normal and 6 = severe inflammation with an overall possible score of 18 points. Higher scores indicate more severe disease. Patients with a total PDAI score >7 points are classed as having pouchitis. The clinical symptom scale assesses stool frequency, rectal bleeding, fecal urgency, and fever. The endoscopic inflammation scale evaluates edema, granularity, friability, loss of vascular pattern, mucus exudates, and ulceration. The modified PDAI is without the histologic findings.

SECONDARY OUTCOMES:
Change from baseline in Simple Endoscopic Score for Crohn's disease (SES-CD) | Baseline and Week 14 and Week 24
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) is a validated tool used to evaluate endoscopic disease activity in Crohn's disease. It assesses four key parameters: (1) the size of ulcers, (2) the ulcerated surface, (3) the affected surface, and (4) the presence of stenosis across five bowel segments (ileum, right colon, transverse colon, left colon, and rectum). Each parameter is scored from 0 to 3 for a total score range of 0-56. Higher scores indicate more severe endoscopic disease activity.
Robarts Histopathology Index (RHI) | Baseline and Week 14 and Week 24
  For histologic assessment, biopsies will be collected and sent for independent central review. Histologic inflammation will be assessed using the Robarts Histopathology Index (RHI) for chronic pouchitis. Each component is scored 0 - 3 and the total possible score is 33, with higher scores reflecting greater histologic disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Phillip Fleshner, M.D. Inc, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No